CLINICAL TRIAL: NCT00860769
Title: ASHA HIV Health Promotion Intervention in India
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Adeline Nyamathi, PhD, Distinguished Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: G071208102; 1 R34 MH082662:01R; 1R34MH082662-01 (NIH)
Record Dates: First submitted 2009-03-11; First posted 2009-03-12 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ASHA Life (Experimental): 6-session educational group discussing HIV prevention, anti-retroviral therapy (ART), coping enhancement, nutrition, parenting and life skills.
  Interventions: Behavioral: ASHA LIFE
- Usual Care (Active Comparator): 3-session educational group focusing on HIV prevention, anti-retroviral therapy (ART) and parenting.
  Interventions: Behavioral: USUAL Care

INTERVENTIONS:
Behavioral: ASHA LIFE — 6-session education groups discussing HIV prevention, anti-retroviral therapy (ART), coping enhancement, nutrition, parenting and life skills
  Arms: ASHA Life
Behavioral: USUAL Care — 3 session educational group focusing on HIV prevention, anti-retroviral therapy and parenting
  Arms: Usual Care

SUMMARY:
The purpose of this randomized pilot study was to conduct an intervention with 68 rural women living with AIDS to compare the effectiveness of two different programs on compliance with HIV/AIDS treatment regimens, improvement in knowledge about HIV/AIDS and TB, improvement in psychological distress, reduction in stigma; satisfaction with care provided to family members, reduction in number of opportunistic infections, increase in CD4 levels and completion of the designed Asha-Life (AL) program. The trial was designed to assess the impact of the Asha-Life (AL) intervention engaging with an HIV-trained village woman, Asha (Accredited Social Health Activist), to participate in the care of women living with AIDS (WLA), along with other health care providers compared to a Usual Care group. Two high prevalence HIV/AIDS villages in rural Andhra Pradesh, which were demographically alike and served by distinct Public Health Centers, were selected randomly from a total of 16 villages.

DETAILED DESCRIPTION:
This Community health study was conducted in two phases:

Phase I was initiated with the establishment of a Community Advisory Board (CAB) composed of 10 persons including WLA, Ashas, and health care providers consisting of Nurse Midwives, HIV and TB experts selected from a Primary Care Clinic in Nellore, Andhra Pradesh. The CAB considered issues related to stigma, disclosure, and psycho-socio-cultural factors affecting the health-seeking behaviors of WLA. They also analyzed the strategies that Asha could employ to support WLA in optimizing their health and well-being and that of their families. This was followed by focus groups conducted separately with the same type of participants. Eligibility criteria included WLA who were currently on ART, were 16-45 years of age, and were able to provide informed consent.

Phase II: A randomized control trial-pilot study was completed in Year 3. We assessed the outcomes of 34 WLA who participated in the AL program at six-month follow-up, as compared with 34 WLA in the Usual Care (UC) Program; in terms of: a) compliance with HIV/AIDS and/or TB treatment regimens (HIV/AIDS/TB), b) improvement in knowledge about HIV/AIDS/TB, c) improvement in psychological distress, d) reduction in stigma, e) reduction in number of opportunistic infections (OIs), f) increase in CD4 levels, and g) completion of the program. The intervention incorporated a comprehensive education and skills program to which we added high protein supplements (1 kg of Black Gram and 1 kg of Toor Dal/month for the AL group vs. a basic program including 1 kg of Channa Dal/month for the UC group.

ELIGIBILITY:
Inclusion Criteria:

* Women living with HIV
* Ages 18-45
* Interfacing with an Accredited Social Health Activist (ASHA)
* Receiving ART or eligible for receiving ART
* HIV Positive status
* CD4 cells ≥ 100
* Not a participant of Phase 1

Exclusion Criteria:

* Cognitively impaired, not a participant of Phase 1

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2008-09; Primary Completion 2011-03 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Conduct a randomized clinical pilot study with 70 women living with HIV in India. | 2 years

SECONDARY OUTCOMES:
Acceptability of the intervention by the women living with HIV. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Adeline Nyamathi, PhD, Principal Investigator — The Regents of the University of California
Locations (1):
- Indian Counsel of Medical Research, New Delhi, India

REFERENCES:
- [Result] Nyamathi A, Ekstrand M, Salem BE, Sinha S, Ganguly KK, Leake B. Impact of Asha intervention on stigma among rural Indian women with AIDS. West J Nurs Res. 2013 Aug;35(7):867-83. doi: 10.1177/0193945913482050. Epub 2013 Mar 27. PMID 23539322
- [Result] Nyamathi A, Hanson AY, Salem BE, Sinha S, Ganguly KK, Leake B, Yadav K, Marfisee M. Impact of a rural village women (Asha) intervention on adherence to antiretroviral therapy in southern India. Nurs Res. 2012 Sep-Oct;61(5):353-62. doi: 10.1097/NNR.0b013e31825fe3ef. PMID 22872107
- [Result] Nyamathi A, Salem BE, Meyer V, Ganguly KK, Sinha S, Ramakrishnan P. Impact of an Asha intervention on depressive symptoms among rural women living with AIDS in India: comparison of the Asha-Life and Usual Care program. AIDS Educ Prev. 2012 Jun;24(3):280-93. doi: 10.1521/aeap.2012.24.3.280. PMID 22676466
- [Result] Nyamathi A, Sinha S, Ganguly KK, Ramakrishna P, Suresh P, Carpenter CL. Impact of protein supplementation and care and support on body composition and CD4 count among HIV-infected women living in rural India: results from a randomized pilot clinical trial. AIDS Behav. 2013 Jul;17(6):2011-21. doi: 10.1007/s10461-013-0420-5. PMID 23370835
- [Result] Nyamathi A, Heravian A, Salem B, Suresh P, Sinha S, Ganguly K, Carpenter C, Ramakrishnan P, Marfisee M, Liu Y. Physical and mental health of rural southern Indian women living with AIDS. J Int Assoc Provid AIDS Care. 2013 Nov-Dec;12(6):391-6. doi: 10.1177/1545109712442241. Epub 2012 May 2. PMID 22553317
- [Result] Nyamathi A, Ekstrand M, Zolt-Gilburne J, Ganguly K, Sinha S, Ramakrishnan P, Suresh P, Marfisee M, Leake B. Correlates of stigma among rural Indian women living with HIV/AIDS. AIDS Behav. 2013 Jan;17(1):329-39. doi: 10.1007/s10461-011-0041-9. PMID 21915715
- [Result] Nyamathi A, Heravian A, Zolt-Gilburne J, Sinha S, Ganguly K, Liu E, Ramakrishnan P, Marfisee M, Leake B. Correlates of depression among rural women living with AIDS in Southern India. Issues Ment Health Nurs. 2011;32(6):385-91. doi: 10.3109/01612840.2011.577269. PMID 21692578
- [Result] Nyamathi AM, Sinha S, Ganguly KK, William RR, Heravian A, Ramakrishnan P, Greengold B, Ekstrand M, Rao PV. Challenges experienced by rural women in India living with AIDS and implications for the delivery of HIV/AIDS care. Health Care Women Int. 2011 Apr;32(4):300-13. doi: 10.1080/07399332.2010.536282. PMID 21409663
- [Result] Nyamathi AM, William RR, Ganguly KK, Sinha S, Heravian A, Albarran CR, Thomas A, Greengold B, Ekstrand M, Ramakrishna P, Rao PR. Perceptions of Women Living with AIDS in Rural India Related to the Engagement of HIV-Trained Accredited Social Health Activists for Care and Support. J HIV AIDS Soc Serv. 2010 Oct;9(4):385-404. doi: 10.1080/15381501.2010.525474. PMID 21331322